CLINICAL TRIAL: NCT00897065
Title: Quantitative Protein and Gene Expression Biomarkers of Tamoxifen and Letrozole Recurrence in the NCIC CTG MA.17 Cohort
Brief Title: Biomarkers in Predicting Response to Tamoxifen and Letrozole in Postmenopausal Women With Primary Breast Cancer Treated on Clinical Trial CAN-NCIC-MA17
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: MGH-MA.17ICSC; CDR0000466578 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2008-04

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Microarray Analysis; Polymerase Chain Reaction; Fluorescent Antibody Technique; Immunohistochemistry; Immunologic Techniques

INTERVENTIONS:
Genetic: microarray analysis
Genetic: polymerase chain reaction
Genetic: protein expression analysis
Other: diagnostic laboratory biomarker analysis
Other: fluorescent antibody technique
Other: immunohistochemistry staining method
Other: immunologic technique

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how well patients respond to treatment.

PURPOSE: This laboratory study is looking at biomarkers that may predict response to tamoxifen and letrozole in postmenopausal women with primary breast cancer treated on clinical trial CAN-NCIC-MA17.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the prognostic utility of the MGH 2-gene and the GHI 21-gene expression signatures in postmenopausal women with primary breast cancer treated with tamoxifen followed by either placebo or letrozole on clinical trial CAN-NCIC-MA17.
* Assess the ability of the MGH 2-gene and the GHI 21-gene expression signatures to predict responsiveness to letrozole.
* Compare the prognostic utility of quantitative immunofluorescence vs standard immunohistochemistry of estrogen receptor, progesterone receptor, HER-2, tumor aromatase, cyclooxygenase-2, GATA-3, and NAT-1 in these patients.
* Assess the ability of quantitative immunofluorescence and standard immunohistochemistry of these proteins to predict responsiveness to letrozole in these patients.
* Use gene discovery from formalin-fixed, paraffin-embedded tumor specimens to identify novel gene expression profiles that may predict outcome and responsiveness to letrozole in these patients.

OUTLINE: This is a controlled study.

Formalin-fixed, paraffin-embedded breast tumor tissue samples are analyzed for MGH 2-gene and GHI 21-gene expression signatures using real-time quantitative polymerase chain reaction. Immunohistochemistry and immunofluorescence are used for analysis of estrogen receptor, progesterone receptor, HER-1 and -2, aromatase, GATA-3, NAT-1, and cyclooxygenase-2. Microarray hybridization is used to identify novel gene expression signatures.

PROJECTED ACCRUAL: A total of 957 specimens will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary invasive breast carcinoma resected at time of original diagnosis
* Treated on clinical trial CAN-NCIC-MA17
* Hormone receptor status:

  * Estrogen or progesterone receptor positive tumor

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 957 (Estimated)
Dates: Start 2006-06

PRIMARY OUTCOMES:
Prognostic utility of the MGH 2-gene and the GHI 21-gene expression signatures
Ability of the MGH 2-gene and the GHI 21-gene expression signatures to predict responsiveness to letrozole
Prognostic utility of quantitative immunofluorescence vs standard immunohistochemistry of estrogen receptor, progesterone receptor, HER-2, tumor aromatase, cyclooxygenase-2, GATA-3, and NAT-1
Ability of quantitative immunofluorescence and standard immunohistochemistry of these proteins to predict responsiveness to letrozole
Novel gene expression profiles that may predict outcome and responsiveness to letrozole

CONTACTS AND LOCATIONS:
Overall Officials: Paul E. Goss, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States